CLINICAL TRIAL: NCT04764604
Title: Evaluating the Therapeutic Use of a Vibratory Positive Expiratory Pressure Device (Acapella® Choice) in the Treatment of Pathological Voice - A Feasibility Study
Brief Title: Evaluating the Feasibility of Acapella® Choice as a Dysphonia Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Smiths Medical, ASD, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/0434
Record Dates: First submitted 2020-11-05; First posted 2021-02-21 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Muscle Tension Dysphonia; Vocal Fold Palsy; Vocal Cord Paralysis; Presbylarynx; Dysphonia
Keywords: semi-occluded vocal tract exercise; positive expiratory pressure; tube phonation; Acapella; voice therapy
MeSH Terms: conditions — Vocal Cord Paralysis; Dysphonia | interventions — Hydrotherapy

STUDY DESIGN:
Intervention Model Description: This is a feasibility study using a 'before and after' design to test the immediate effects of exercising with Acapella Choice in comparison to the immediate effects of exercising with Tube-in-water resistance exercises (current treatment norm). Participants will be assigned groups according to their diagnosis (i.e. muscle tension group, vocal fold palsy group and presbylaryngis group). All participants will exercise with both techniques (i.e. Acapella and tube-in-water).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Muscle Tension Group (Experimental): 10 participants with a diagnosis of muscle tension dysphonia will carry out two experimental interventions, with a 30 minute vocal rest period in between interventions:
  1. Three minutes of semi-occluded vocal tract exercise with both Acapella Choice
  2. Three minutes of tube-in-water semi-occluded vocal tract exercise.
  Aerodynamic, acoustic and electroglottographic baselines will be taken before each intervention and repeated immediately post-intervention as outcomes.
  Participants will also provide a self-assessment of voice quality, perceived ease of voice production and perceived strength of voice before and after each intervention.
  Participants will additionally answer qualitative questions following each intervention regarding their perceptions of the task: ease performing, pleasantness, effort, practicality and likelihood of carrying out the task on a daily basis as a form of therapy.
  Interventions: Device: Acapella Choice; Device: Tube-in-water
- Vocal Fold Palsy Group (Experimental): 10 participants with a diagnosis of (unilateral) vocal fold palsy will carry out two experimental interventions, with a 30 minute vocal rest period in between interventions:
  1. Three minutes of semi-occluded vocal tract exercise with both Acapella Choice
  2. Three minutes of tube-in-water semi-occluded vocal tract exercise.
  Aerodynamic, acoustic and electroglottographic baselines will be taken before each intervention and repeated immediately post-intervention as outcomes.
  Participants will also provide a self-assessment of voice quality, perceived ease of voice production and perceived strength of voice before and after each intervention.
  Participants will additionally answer qualitative questions following each intervention regarding their perceptions of the task: ease performing, pleasantness, effort, practicality and likelihood of carrying out the task on a daily basis as a form of therapy.
  Interventions: Device: Acapella Choice; Device: Tube-in-water
- Presbylaryngis Group (Experimental): 10 participants with a diagnosis of presbylaryngis will carry out two experimental interventions, with a 30 minute vocal rest period in between interventions:
  1. Three minutes of semi-occluded vocal tract exercise with both Acapella Choice
  2. Three minutes of tube-in-water semi-occluded vocal tract exercise.
  Aerodynamic, acoustic and electroglottographic baselines will be taken before each intervention and repeated immediately post-intervention as outcomes.
  Participants will also provide a self-assessment of voice quality, perceived ease of voice production and perceived strength of voice before and after each intervention.
  Participants will additionally answer qualitative questions following each intervention regarding their perceptions of the task: ease performing, pleasantness, effort, practicality and likelihood of carrying out the task on a daily basis as a form of therapy.
  Interventions: Device: Acapella Choice; Device: Tube-in-water

INTERVENTIONS:
Device: Acapella Choice — 3 minutes of exercise consisting of blowing through the device (on setting '5') and phonating at the same time.
  Other Names: PEP; Semioccluded vocal tract exercise
Device: Tube-in-water — 3 minutes of exercise consisting of blowing through a silicone tube (10mm internal diameter) submerged in 5 cm of water whilst phonating at the same time.
  Other Names: Lax Vox; Resonance tube in water; Semi-occluded vocal tract exercise

SUMMARY:
A feasibility study to identify the immediate effect on the voices of patients with voice disorders (muscle tension dysphonia, vocal fold palsy or presbylaryngis) produced by exercising with Acapella Choice as a form of semioccluded vocal tract exercise (SOVTE).

DETAILED DESCRIPTION:
This feasibility study is the natural extension of the researchers' recently completed study (R&D 16/0242) which assessed how the use of an Acapella Choice (Smiths Medical) positive expiratory pressure (PEP) device as a semi-occluded vocal tract exercise (SOVTE) impacted acoustic, electroglottographic and aerodynamic measures of the voice in a group of normophonic volunteers. In that study, Acapella Choice was found to offer significantly greater oscillating intraoral pressures than techniques in current clinical practice and was found to have measurable benefits in terms of producing a louder and more economical voice. It offered the largest oscillating pressures, likened to a 'massage' of the vocal organs, giving it great therapeutic promise for patients with excess vocal tract tension.

This study seeks to evaluate the immediate effects of Acapella Choice as a voice exercise in patients with Muscle Tension Dysphonia, Presbylaryngis and Vocal Fold Palsy, and compare this to the widely-used voice rehabilitation technique of phonation into a tube held under water (henceforward referred to as "Tube"). Patients will be recruited from four weekly Voice Clinics held at the Royal National Throat Nose and Ear Hospital where their diagnosis will be confirmed. They will be invited to attend a single experimental session during which time they will exercise both with Acapella Choice and with Tube. Baseline and outcome voice measures will be taken and a short questionnaire will be completed, eliciting perceptions of the two exercises and any changes which were felt to have resulted from them.

The researchers' previous work suggests that Acapella Choice as a SOVTE may offer significant clinical benefits in terms of improved efficacy of therapy. It is suggested that it also offers patients a more convenient and user-friendly form of exercise which may well improve compliance and result in better outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand written English without the need for an interpreter,
* No diagnosed communication impairment
* Endoscopically confirmed primary ENT diagnosis of either:

  1. muscle tension dysphonia (with no laryngeal abnormality),
  2. Vocal fold palsy
  3. Presbylaryngis.

Exclusion Criteria:

* Previous SLT input
* Any of the following possible contraindications for PEP therapy:

  * Inability to tolerate increased work of breathing,
  * ICP (intracranial pressure) > 20mm Hg,
  * Recent facial/oral/skull surgery or trauma,
  * Oesophageal surgery,
  * Untreated pneumothorax,
  * Known or suspected tympanic membrane rupture/other middle ear pathology,
  * Haemodynamic instability,
  * Acute sinusitis,
  * Epistaxis,
  * Active haemoptysis,
  * Nausea

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Saccente-Kennedy, MSc, Principal Investigator — University College London Hospitals
Locations (1):
- Royal National ENT Hospital, UCLH Hospitals NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Titze IR, Story BH. Acoustic interactions of the voice source with the lower vocal tract. J Acoust Soc Am. 1997 Apr;101(4):2234-43. doi: 10.1121/1.418246. PMID 9104025
- [Background] Titze IR. Voice training and therapy with a semi-occluded vocal tract: rationale and scientific underpinnings. J Speech Lang Hear Res. 2006 Apr;49(2):448-59. doi: 10.1044/1092-4388(2006/035). PMID 16671856
- [Background] Sovijärvi A. Die Bestimmung der Stimmkategorien mittels Resonanzröhren. [Voice classification according to resonance tubes]. In: Fifth International Congress of Phonetic Sciences. Basel, NY. ; 1965.
- [Background] Simberg S, Laine A. The resonance tube method in voice therapy: description and practical implementations. Logoped Phoniatr Vocol. 2007;32(4):165-70. doi: 10.1080/14015430701207790. PMID 17852715
- [Background] Enflo L, Sundberg J, Romedahl C, McAllister A. Effects on vocal fold collision and phonation threshold pressure of resonance tube phonation with tube end in water. J Speech Lang Hear Res. 2013 Oct;56(5):1530-8. doi: 10.1044/1092-4388(2013/12-0040). Epub 2013 Jul 9. PMID 23838993
- [Background] Granqvist S, Simberg S, Hertegard S, Holmqvist S, Larsson H, Lindestad PA, Sodersten M, Hammarberg B. Resonance tube phonation in water: High-speed imaging, electroglottographic and oral pressure observations of vocal fold vibrations--a pilot study. Logoped Phoniatr Vocol. 2015 Oct;40(3):113-21. doi: 10.3109/14015439.2014.913682. Epub 2014 May 28. PMID 24865620
- [Background] Wistbacka G, Sundberg J, Simberg S. Vertical laryngeal position and oral pressure variations during resonance tube phonation in water and in air. A pilot study. Logoped Phoniatr Vocol. 2016 Oct;41(3):117-23. doi: 10.3109/14015439.2015.1028101. Epub 2015 Jun 2. PMID 26033381
- [Background] Amarante Andrade P, Wistbacka G, Larsson H, Sodersten M, Hammarberg B, Simberg S, Svec JG, Granqvist S. The Flow and Pressure Relationships in Different Tubes Commonly Used for Semi-occluded Vocal Tract Exercises. J Voice. 2016 Jan;30(1):36-41. doi: 10.1016/j.jvoice.2015.02.004. Epub 2015 Apr 11. PMID 25873546
- [Background] Andrade PA, Wood G, Ratcliffe P, Epstein R, Pijper A, Svec JG. Electroglottographic study of seven semi-occluded exercises: LaxVox, straw, lip-trill, tongue-trill, humming, hand-over-mouth, and tongue-trill combined with hand-over-mouth. J Voice. 2014 Sep;28(5):589-95. doi: 10.1016/j.jvoice.2013.11.004. Epub 2014 Feb 20. PMID 24560003
- [Background] Guzman M, Castro C, Madrid S, Olavarria C, Leiva M, Munoz D, Jaramillo E, Laukkanen AM. Air Pressure and Contact Quotient Measures During Different Semioccluded Postures in Subjects With Different Voice Conditions. J Voice. 2016 Nov;30(6):759.e1-759.e10. doi: 10.1016/j.jvoice.2015.09.010. Epub 2016 Jun 13. PMID 26526005
- [Background] Radolf V, Laukkanen A, Horacek J, Liu D. In vivo measurements of air pressure, vocal folds vibration and acoustic characteristics of phonation into a straw and resonance tube used in vocal exercising. In: Proceedings of the 19th International Conference Engineering Mechanics, Czech Republic. ; 2013:478-483.
- [Background] Awan SN, Gartner-Schmidt JL, Timmons LK, Gillespie AI. Effects of a Variably Occluded Face Mask on the Aerodynamic and Acoustic Characteristics of Connected Speech in Patients With and Without Voice Disorders. J Voice. 2019 Sep;33(5):809.e1-809.e10. doi: 10.1016/j.jvoice.2018.03.002. Epub 2018 Aug 3. PMID 30082107
- [Background] Guzman M, Calvache C, Romero L, Munoz D, Olavarria C, Madrid S, Leiva M, Bortnem C, Pino J. Do Different Semi-Occluded Voice Exercises Affect Vocal Fold Adduction Differently in Subjects Diagnosed with Hyperfunctional Dysphonia? Folia Phoniatr Logop. 2015;67(2):68-75. doi: 10.1159/000437353. Epub 2015 Sep 23. PMID 26394210
- [Background] Guzman M, Higueras D, Fincheira C, Munoz D, Guajardo C, Dowdall J. Immediate acoustic effects of straw phonation exercises in subjects with dysphonic voices. Logoped Phoniatr Vocol. 2013 Apr;38(1):35-45. doi: 10.3109/14015439.2012.731079. Epub 2013 Jan 28. PMID 23350916
- [Background] Guzman M, Laukkanen AM, Krupa P, Horacek J, Svec JG, Geneid A. Vocal tract and glottal function during and after vocal exercising with resonance tube and straw. J Voice. 2013 Jul;27(4):523.e19-34. doi: 10.1016/j.jvoice.2013.02.007. Epub 2013 May 15. PMID 23683806
- [Background] Gaskill CS, Erickson ML. The effect of a voiced lip trill on estimated glottal closed quotient. J Voice. 2008 Nov;22(6):634-43. doi: 10.1016/j.jvoice.2007.03.012. Epub 2007 Jun 15. PMID 17574810
- [Background] Gaskill CS, Quinney DM. The effect of resonance tubes on glottal contact quotient with and without task instruction: a comparison of trained and untrained voices. J Voice. 2012 May;26(3):e79-93. doi: 10.1016/j.jvoice.2011.03.003. Epub 2011 May 7. PMID 21550779
- [Background] Gaskill CS, Erickson ML. The effect of an artificially lengthened vocal tract on estimated glottal contact quotient in untrained male voices. J Voice. 2010 Jan;24(1):57-71. doi: 10.1016/j.jvoice.2008.05.004. Epub 2009 Jan 9. PMID 19135851
- [Background] Guzman M, Castro C, Testart A, Munoz D, Gerhard J. Laryngeal and pharyngeal activity during semioccluded vocal tract postures in subjects diagnosed with hyperfunctional dysphonia. J Voice. 2013 Nov;27(6):709-16. doi: 10.1016/j.jvoice.2013.05.007. Epub 2013 Sep 26. PMID 24075912
- [Background] Vampola T, Laukkanen AM, Horacek J, Svec JG. Vocal tract changes caused by phonation into a tube: a case study using computer tomography and finite-element modeling. J Acoust Soc Am. 2011 Jan;129(1):310-5. doi: 10.1121/1.3506347. PMID 21303012
- [Background] Patterson JE, Hewitt O, Kent L, Bradbury I, Elborn JS, Bradley JM. Acapella versus 'usual airway clearance' during acute exacerbation in bronchiectasis: a randomized crossover trial. Chron Respir Dis. 2007;4(2):67-74. doi: 10.1177/1479972306075483. PMID 17621572
- [Background] Mueller G, Bersch-Porada I, Koch-Borner S, Raab AM, Jonker M, Baumberger M, Michel F. Laboratory evaluation of four different devices for secretion mobilization: Acapella choice, green and blue versus water bottle. Respir Care. 2014 May;59(5):673-7. doi: 10.4187/respcare.02654. Epub 2013 Sep 17. PMID 24046459

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Laryngeal Resistance: Recruited participants will be stratified into Low and High Laryngeal Resistance Groups on the basis of their baseline (i.e. before intervention) laryngeal resistance as compared to published norms. Laryngeal resistance is derived from dividing mean intraoral pressure (in cmH2O) during /p/ by mean transglottic airflow (in l/s) during /a/ during a task which elicits repetition of 'pa-pa-pa-pa-pa'. This resistance will then be converted into a Z-score in relation to published norms. Those participants with a laryngeal resistance below a Z-score of 0 (i.e age- and gender-matched published normative mean) will be categorised into the 'low laryngeal resistance group'.
  All participants will perform the following tasks:
  1. Three minutes of semi-occluded vocal tract exercise with both Acapella Choice
  2. Three minutes of tube-in-water semi-occluded vocal tract exercise.
  Aerodynamic, acoustic and electroglottographic baselines will be taken before each intervention and repeated immediately post-intervention as outcomes.
  Participants will also provide a self-assessment of voice quality, perceived ease of voice production and perceived strength of voice before and after each intervention.
  Participants will additionally answer qualitative questions following each intervention regarding their perceptions of the task: ease performing, pleasantness, effort, practicality and likelihood of carrying out the task on a daily basis as a form of therapy.
- High Laryngeal Resistance Group: Recruited participants will be stratified into Low and High Laryngeal Resistance Groups on the basis of their baseline (i.e. before intervention) laryngeal resistance as compared to published norms. Laryngeal resistance is derived from dividing mean intraoral pressure (in cmH2O) during /p/ by mean transglottic airflow (in l/s) during /a/ during a task which elicits repetition of 'pa-pa-pa-pa-pa'. This resistance will then be converted into a Z-score in relation to published norms. Those participants with a laryngeal resistance above a Z-score of 0 (i.e age- and gender-matched published normative mean) will be categorised into the 'high laryngeal resistance group'.
  All participants will perform the following tasks:
  1. Three minutes of semi-occluded vocal tract exercise with both Acapella Choice
  2. Three minutes of tube-in-water semi-occluded vocal tract exercise.
  Aerodynamic, acoustic and electroglottographic baselines will be taken before each intervention and repeated immediately post-intervention as outcomes.
  Participants will also provide a self-assessment of voice quality, perceived ease of voice production and perceived strength of voice before and after each intervention.
  Participants will additionally answer qualitative questions following each intervention regarding their perceptions of the task: ease performing, pleasantness, effort, practicality and likelihood of carrying out the task on a daily basis as a form of therapy.
Period: Overall Study
Arm/Group | Low Laryngeal Resistance | High Laryngeal Resistance Group
Started | 16 | 14
Acapella Choice Task | 16 | 14
Tube-in-Water Task | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Recruitment was undertaken along the lines of laryngeal diagnosis (10 patients in each diagnosis category). However, as laryngeal diagnosis results in diverse behavioural responses, treatment is never determined by diagnosis, alone. To better understand how participants responded to treatment, they were stratified into meaningful functional categories (Low and High Laryngeal Resistance), as these better represent the physiological targets of voice therapy.
Groups:
- Low Laryngeal Resistance: N=14. Laryngeal resistance with Z-scores for laryngeal resistance below 0.
- High Laryngeal Resistance: N=16. Laryngeal resistance with Z-scores for laryngeal resistance above 0.
- Total: Total of all reporting groups
Arm/Group | Low Laryngeal Resistance | High Laryngeal Resistance | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.31 (16.8) | 58.14 (18.9) | 55.0 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 6 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16 | 14 | 30
Aerodynamic Resistance (Z-score) [Median (Inter-Quartile Range); unit: Z scores] — Laryngeal resistance (subglottic pressure divided by transglottic airflow) is known to vary by age and gender. As such, participant aerodynamic resistance was converted to a Z-score in relation to published age and gender-based norms to account for normal variability between participants. The Z-score central value (0) represents the published population mean. Both abnormally high and abnormally low laryngeal resistance would reflect disordered laryngeal function in phonation (in this case strained vs overly breathy phonation). Clinically meaningful thresholds have not been established.
  Z scores | -0.63 [-1.09 to -0.18] | 1.07 [-0.16 to 2.30] | -0.21 [-0.81 to 0.39]

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline Cepstral/Spectral Index of Dysphonia (CSID)
Description: A quantitative, multivariate, dysphonia summary tool that incorporates spectral (low/high spectral ratio) and cepstral measures (cepstral peak prominence), and their standard deviations, extracted from a continuous speech or sustained vowel sample utilising the software Analysis of Dysphonia in Speech and Voice (Kay Pentax, Montvale, NJ). The software calculates CSID on the scale of 0-100, whereby 0 represents no evidence of hoarse voice, and 100 represents a maximum amount of hoarseness. See: Awan SN, Roy N, Dromey C. Estimating dysphonia severity in continuous speech: Application of a multi-parameter spectralcepstral model estimating dysphonia severity in continuous speech. Clinical Linguistics and Phonetics. 2009;23(11):825-841. doi:10.3109/02699200903242988.
Time Frame: Immediately after 3 minutes of exercise
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Laryngeal Resistance | High Laryngeal Resistance
Number analyzed (Participants) | 14 | 16
score on a scale
  Acapella Task | 1.22 (7.72) | 4.45 (12.2)
  WRT Task | 4.56 (13.1) | 3.13 (8.21)

2. Secondary Outcome: Change in Baseline Sound Pressure Level (dB)
Description: Intensity of vocal signal
Time Frame: Immediately after 3 minutes of exercise
Population: Each subgroup (Low and High Laryngeal Resistance) underwent two therapeutic interventions (Acapella and Water Resistance Therapy (WRT)) each.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Low Laryngeal Resistance | High Laryngeal Resistance
Number analyzed (Participants) | 14 | 16
dB
  Acapella Task | 0.79 (1.97) | 1.46 (2.72)
  WRT Task | 1.57 (2.98) | -0.52 (2.76)

3. Secondary Outcome: Change in Baseline Mean Contact Quotient
Description: A percentage which illustrates the duration of vocal fold contact during one vocal fold period as measured by electroglottogram (EGG).
Time Frame: During 3 minutes of exercise (continual) and immediately following exercise.
Measure: Mean (Standard Deviation); unit: percentage of contact
Arm/Group | Low Laryngeal Resistance | High Laryngeal Resistance
Number analyzed (Participants) | 14 | 16
percentage of contact
  Acapella Task | 0.01 (0.04) | -0.01 (0.06)
  WRT Task | 0.01 (0.06) | 0.00 (0.03)

4. Secondary Outcome: Change in Subglottic Pressure
Description: Measures of air pressure in the mouth.
Time Frame: During 3 minutes of exercise (continual)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Low Laryngeal Resistance | High Laryngeal Resistance
Number analyzed (Participants) | 14 | 16
cmH2O
  Acapella Task | 0.16 (1.72) | 0.95 (1.81)
  WRT Task | -0.74 (0.61) | -0.68 (1.77)

5. Secondary Outcome: Transglottic Airflow
Description: Measures of flow of air through the vocal tract.
Time Frame: During 3 minutes of exercise (continual)
Measure: Mean (Standard Deviation); unit: l/s
Arm/Group | Low Laryngeal Resistance | High Laryngeal Resistance
Number analyzed (Participants) | 14 | 16
l/s
  Acapella Task | 0.017 (0.163) | 0.023 (0.075)
  WRT Task | -0.011 (0.097) | -0.003 (0.061)

6. Secondary Outcome: Change in Baseline Laryngeal Resistance
Description: Derived from dividing mean intraoral pressure during /p/ by mean transglottic airflow during /a/ during a task which elicits repetition of 'pa-pa-pa-pa-pa'
Time Frame: Immediately after 3 minutes of exercise
Population: In this outcome, pre-port comparison is made with actual units of resistance. Previously, Z-scores were utilised to explain the baseline differences between the groups (i.e. low vs high resistance groups). In the case of this outcome measure, a per-participant difference in pre- and post-exercise resistance is utilised.
Measure: Mean (Standard Deviation); unit: cmH20/l/s
Arm/Group | Low Laryngeal Resistance | High Laryngeal Resistance
Number analyzed (Participants) | 14 | 16
cmH20/l/s
  Acapella Task | 1.40 (23.9) | -6.01 (58.7)
  WRT Task | -5.04 (14.5) | 23.77 (122)

7. Secondary Outcome: Change in Baseline Perceptual Voice Quality
Description: Expert ratings of overall voice quality using a simple ad-hoc 100mm visual analog scale (ranging from 0-100, reflecting a scale of normal voice quality to highly abnormal voice quality {higher numbers reflect more abnormality}).
Time Frame: Immediately after 3 minutes of exercise
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Laryngeal Resistance | High Laryngeal Resistance
Number analyzed (Participants) | 14 | 16
units on a scale
  Acapella Task | -1.82 (6.03) | 0.175 (4.73)
  WRT Task | 0.622 (4.65) | 5.18 (4.92)

8. Secondary Outcome: Change in Baseline Participant Self-ratings - Voice Quality
Description: Participant self-rating of voice quality (on a 100mm visual analog scale (0-100) where higher numbers reflect self-perception of better voice quality/ease of production)
Time Frame: Immediately after 3 minutes of exercise
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Laryngeal Resistance | High Laryngeal Resistance
Number analyzed (Participants) | 14 | 16
units on a scale
  Acapella Task | 12.3 (13.8) | 4.62 (9.05)
  WRT Task | 6.56 (11.1) | 1.38 (9.97)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Low Laryngeal Resistance | High Laryngeal Resistance
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT04764604/Prot_SAP_000.pdf